CLINICAL TRIAL: NCT03194490
Title: Benefit of Adding Stretching to Standard Intervention For Patients With Nonspecific Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Everett Lohman, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5160230
Record Dates: First submitted 2017-06-13; First posted 2017-06-21 (Actual); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The combined intervention group (Experimental): The combined intervention group will receive the cervical passive mobilization, stretching, and home program (Stretching and ROM exercise).
  Interventions: Other: combined intervention group
- The standard intervention (Active Comparator): The standard intervention group will receive cervical mobilization and home program (ROM exercises).
  Interventions: Other: The standard intervention

INTERVENTIONS:
Other: combined intervention group — The combined intervention group received the cervical passive mobilization, stretching, and home program (Stretching and ROM exercise).Stretching, cervical passive mobilization, and range of motion: The manual therapy was conducted by a physical therapist who has licensed from the California Board of Physical Therapy. The cervical passive mobilization were selected by the physical therapist based on the participant's condition. Stretching techniques were performed in the combined intervention group for 30 seconds and repeated 3 times twice a week in the following order on the following muscles: anterior, middle and posterior scalene, upper fibers of trapezius, pectoralis minor and interspinous muscles .AROM Exercise were performed 10 repetitions 3-4 times daily. The ACROM exercise consisted of the subject placing fingers over the manubrium bone and placing chin on the fingers. The subject was then instructed to rotate to one side as far as possible and return to neutral.
  Arms: The combined intervention group
Other: The standard intervention — The standard intervention group will receive cervical mobilization and home program (ROM exercises).
  Cervical mobilization and range of motion: The manual therapy was conducted by a physical therapist who has experience in manual therapy and is licensed from the California Board of Physical Therapy. The manual therapy intervention will consist of Passive Accessory Intervertebral Movements (PAIVMs). The nature of PAIVMs techniques was selected by the physical therapist based on the participant's condition.
  Active Cervical Range of Motion Exercises (ACROM) were performed 10 repetitions 3-4 times daily. Subjects were advised to maintain their usual activity within the limits of pain. The ACROM exercise consisted of the subject placing fingers over the manubrium bone and placing chin on the fingers. The subject was then instructed to rotate to one side as far as possible and return to neutral .
  Arms: The standard intervention

SUMMARY:
The purpose of this study is to assess the benefit of adding stretching exercises to cervical mobilization and cervical range of motion exercises on cervical range of motion, pain, pain threshold, level of disability and patient satisfaction for patient with non-specific mechanical neck pain

DETAILED DESCRIPTION:
All recruited participants will sign a statement of informed consent. Subjects were randomly divided into two groups (combined intervention group and standard intervention group). The following questionnaires were completed in the following order: Neck Disability Index (NDI), Numeric Pain Rating Scale (NPRS), and Global Rating of Change Scale (GROC). Next, Cervical Range of Motion (ROM) and Pain threshold were measured for both groups. The combined intervention group received the cervical passive mobilization, stretching, and home program (Stretching and ROM exercise). The standard intervention group received cervical mobilization and home program (ROM exercises).

ELIGIBILITY:
Inclusion Criteria:

* The participant will be eligible to participate in the study if he or she is between 18 and 60 years of age, had non-specific neck pain for at least 2 weeks

Exclusion Criteria:

* Participants will be excluded from the study if they had one or more of the following conditions: had previous surgery in cervical spine area, chronic disease such as diabetes, vertigo, dizziness, fracture of the cervical vertebra or scapula, multiple sclerosis, osteoporosis, rheumatoid arthritis or osteoarthritis as approximately 60% of people who aged between 50-60 years will have osteoarthritis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett B Lohman, Principal Investigator — Loma Linda U
Locations (1):
- Loma Linda U, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Intervention Group: The combined intervention group received the cervical passive mobilization, stretching, and home program (Stretching and ROM exercise).
  Stretching, cervical passive mobilization, and range of motion: The manual therapy was conducted by a physical therapist who has experience in manual therapy and is licensed from the California Board of Physical Therapy. The manual therapy intervention will consist of Passive Accessory Intervertebral Movements (PAIVMs). The nature of PAIVMs techniques were selected by the physical therapist based on the participant's condition.
  Stretching exercise will be given to the participants by the physical therapist. Stretching techniques were performed in the combined intervention group for 30 seconds and repeated 3 times twice a week in the following order on the following muscles: anterior, middle and posterior scalene, upper fibers of trapezius, pectoralis minor muscles and interspinous muscles.
- The Standard Intervention: The standard intervention group will receive cervical mobilization and home program (ROM exercises).
  Cervical mobilization and range of motion: The manual therapy was conducted by a physical therapist who has experience in manual therapy and is licensed from the California Board of Physical Therapy. The manual therapy intervention will consist of Passive Accessory Intervertebral Movements (PAIVMs). The nature of PAIVMs techniques was selected by the physical therapist based on the participant's condition.
  Active Cervical Range of Motion Exercises (ACROM) were performed 10 repetitions 3-4 times daily. Subjects were advised to maintain their usual activity within the limits of pain. The ACROM exercise consisted of the subject placing fingers over the manubrium bone and placing chin on the fingers. The subject was then instructed to rotate to one side as far as possible and return to neutral.
Period: Overall Study
Arm/Group | Combined Intervention Group | The Standard Intervention
Started | 20 | 23
Completed | 18 | 20
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 3
Not completed — participant developed specific neck pain | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- The Combined Intervention Group: The combined intervention group: The combined intervention group received the cervical passive mobilization, stretching, and home program (Stretching and ROM exercise).
  Stretching, cervical passive mobilization, and range of motion: The manual therapy was conducted by a physical therapist who has experience in manual therapy and is licensed from the California Board of Physical Therapy. The manual therapy intervention will consist of Passive Accessory Intervertebral Movements (PAIVMs). The nature of PAIVMs techniques were selected by the physical therapist based on the participant's condition.
  Stretching exercise will be given to the participants by the physical therapist. Stretching techniques were performed in the combined intervention group for 30 seconds and repeated 3 times twice a week in the following order on the following muscles: anterior, middle and posterior scalene, upper fibers of trapezius, pectoralis minor muscles and interspinous muscles.
- The Standard Intervention: The standard intervention: The standard intervention group received cervical mobilization and home program (ROM exercises).
  Cervical mobilization and range of motion: The manual therapy was conducted by a physical therapist who has experience in manual therapy and is licensed from the California Board of Physical Therapy. The manual therapy intervention will consist of Passive Accessory Intervertebral Movements (PAIVMs). The nature of PAIVMs techniques was selected by the physical therapist based on the participant's condition.
  Active Cervical Range of Motion Exercises (ACROM) were performed 10 repetitions 3-4 times daily. Subjects were advised to maintain their usual activity within the limits of pain. The ACROM exercise consisted of the subject placing fingers over the manubrium bone and placing chin on the fingers. The subject was then instructed to rotate to one side as far as possible and return to neutral.
- Total: Total of all reporting groups
Arm/Group | The Combined Intervention Group | The Standard Intervention | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 38
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (9.0) | 30.6 (7.8) | 31 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 18 | 20 | 38
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 38

OUTCOME MEASURES:

1. Primary Outcome: Cervical Range of Motion
Description: The cervical range of motion device (CROM) will be used to assess the changes in active range of motion for cervical rotation, flexion and extension when comparing baseline,week two, four and eight.
Time Frame: Participants ROM measurement at baselines
Measure: Mean (Standard Error); unit: Degree
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Degree
  Flexion | 46.2 (2.6) | 46.1 (2.2)
  Extesion | 71.2 (3.4) | 68.5 (2.4)
  Right Rotation | 65.9 (3.0) | 66.1 (2.5)
  Left Rotation | 60.1 (3.8) | 62.7 (2.1)
  Right Lateral Flexion | 41.8 (2.5) | 39.9 (1.9)
  Left Lateral Flexion | 43.9 (1.9) | 42.2 (1.4)

2. Primary Outcome: Cervical Range of Motion
Description: The cervical range of motion device (CROM) will be used to assess the changes in active range of motion for cervical rotation, flexion and extension when comparing baseline, week two, four and eight.
Time Frame: Participants ROM measurement at week 2
Measure: Mean (Standard Error); unit: Degree
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Degree
  Flexion | 52.3 (2.4) | 49.7 (2.3)
  Extesion | 77.5 (2.7) | 71.1 (3.7)
  Right Rotation | 71.9 (3.1) | 68.6 (2.4)
  Left Rotation | 66.8 (2.6) | 67.8 (2.1)
  Right Lateral Flexion | 46.3 (1.7) | 41.3 (2.0)
  Left Lateral Flexion | 48.4 (1.6) | 44.3 (1.3)

3. Primary Outcome: Cervical Range of Motion
Description: as for outcome 2
Time Frame: Participants measurement at week four
Measure: Mean (Standard Error); unit: Degree
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Degree
  Flexion | 54.9 (2.5) | 55.0 (2.3)
  Extesion | 82.9 (3.1) | 70.3 (3.1)
  Right Rotation | 74.0 (3.4) | 74.3 (2.5)
  Left Rotation | 73.0 (2.2) | 70.6 (2.3)
  Right Lateral Flexion | 50.0 (2.1) | 43.6 (1.8)
  Left Lateral Flexion | 51.6 (2.1) | 45.3 (1.6)

4. Primary Outcome: Cervical Range of Motion
Description: as for outcome 1
Time Frame: Participants ROM measurement at week 8
Measure: Mean (Standard Error); unit: Degree
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Degree
  Flexion | 53.9 (2.5) | 53.2 (2.6)
  Extesion | 79.2 (2.8) | 74.5 (4.0)
  Right Rotation | 78.5 (2.5) | 71.5 (2.8)
  Left Rotation | 72.9 (2.4) | 71.3 (2.1)
  Right Lateral Flexion | 51.2 (2.4) | 47.3 (1.9)
  Left Lateral Flexion | 55.3 (2.6) | 74.4 (1.9)

5. Secondary Outcome: Numeric Pain Rating Scale
Description: Numeric pain rating scale (NPRS) is a liner outcome measurement used to determine the level of the participant's pain when comparing baseline, week two, four and eight. It consists of a straight 10 cm line that is scored from 0 to 10 with 10 mm intervals. The zero represents no pain while a 10 represents very severe pain that participant cannot stand. The standard error is correct as stated.
Time Frame: NPRS score at baseline
Measure: Mean (Standard Error); unit: Cm
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Cm | 5.2 (0.4) | 4.3 (0.4)

6. Secondary Outcome: Numeric Pain Rating Scale
Description: Numeric pain rating scale (NPRS) is a liner outcome measurement used to determine the level of the participant's pain when comparing baseline, week two, four and eight. It consists of a straight 10 cm line that is scored from 0 to 10 with 10 mm intervals. The zero represents no pain while a 10 represents very severe pain that participant cannot stand.
Time Frame: NPRS score at week two
Measure: Mean (Standard Error); unit: Cm
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Cm | 3.6 (0.4) | 3.0 (0.4)

7. Secondary Outcome: Numeric Pain Rating Scale
Description: as for outcome 6
Time Frame: NPRS score at week four
Measure: Mean (Standard Error); unit: Cm
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Cm | 1.7 (0.4) | 1.8 (0.4)

8. Secondary Outcome: Numeric Pain Rating Scale
Description: as for outcome 6
Time Frame: NPRS score at week eight
Measure: Mean (Standard Error); unit: Cm
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
Cm | 1.5 (0.5) | 1.8 (0.6)

9. Secondary Outcome: Neck Disability Index
Description: Neck disability index measuring the level of neck disability when comparing baseline, week two, four, and eight. It consists of ten items each item is scored from 0 to 5 with a minimum score 0 and highest score 50. A score of zero (0) represents no disability while a score of 50 represents severe, full disability.
Time Frame: NDI score at baseline
Measure: Mean (Standard Error); unit: points
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
points | 12.2 (1.1) | 10.6 (1.1)

10. Secondary Outcome: Neck Disability Index
Description: as for outcome 9
Time Frame: NDI score at week two
Measure: Mean (Standard Error); unit: points
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
points | 7.2 (1.0) | 8.1 (0.9)

11. Secondary Outcome: Neck Disability Index
Description: as for outcome 9
Time Frame: NDI score at week four
Measure: Mean (Standard Error); unit: points
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
points | 3.8 (1.2) | 5.1 (1.1)

12. Secondary Outcome: Neck Disability Index
Description: as for outcome 9
Time Frame: NDI score at week eight
Measure: Mean (Standard Error); unit: points
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
points | 3.7 (1.0) | 6.5 (2.6)

13. Secondary Outcome: Global Rating of Change
Description: The Global rating of change (GROC) is used to measure the amount of improvement that the patient achieves from the intervention or rehabilitation program when comparing baseline, week two, four, and eight. The score ranges from -7 to 0 to 7 in which -/+3 to -/+ 1 represents a small change, -/+ 4 to -/+5 represents moderate change and -/+6 to -/+7 means a large change. The negative and positive means the patient condition worsens or improves respectively. The points are scores on a scale (-7-0-+7 = 15 point scale).
Time Frame: GROC score at week two
Measure: Mean (Standard Error); unit: points
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
points | 2.6 (0.5) | 2.1 (0.5)

14. Secondary Outcome: Global Rating of Change
Description: The Global rating of change (GROC) is used to measure the amount of improvement that the patient achieves from the intervention or rehabilitation program when comparing baseline, week two, four and eight. The score ranges from -7 to 0 to 7 in which -/+3 to -/+ 1 represents a small change, -/+ 4 to -/+5 represents moderate change and -/+6 to -/+7 means a large change. The negative and positive means the patient condition worsens or improves respectively.
Time Frame: GROC score at week four
Measure: Mean (Standard Error); unit: points
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
points | 4.9 (0.5) | 4.5 (0.5)

15. Secondary Outcome: Global Rating of Change
Description: The Global rating of change (GROC) is used to measure the amount of improvement that the patient achieves from the intervention or rehabilitation program when comparing baseline, week two, four and right. The score ranges from -7 to 0 to 7 in which -/+3 to -/+ 1 represents a small change, -/+ 4 to -/+5 represents moderate change and -/+6 to -/+7 means a large change. The negative and positive means the patient condition worsens or improves respectively.
Time Frame: GROC score at week eight
Measure: Mean (Standard Error); unit: points
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
points | 4.9 (0.6) | 3.3 (1.0)

16. Secondary Outcome: Pressure Pain Threshold
Description: Pressure pain threshold is an electronic device used to measure the amount of force that is required to produce pain when comparing baseline, week two, four, and eight.
Time Frame: Pressure Pain Threshold score at baseline
Measure: Mean (Standard Error); unit: pound per centimeter square
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
pound per centimeter square
  Right Pressure Pain Threshold | 4.5 (0.4) | 5.0 (0.5)
  Left Pressure Pain Threshold | 4.3 (0.4) | 4.7 (0.4)

17. Secondary Outcome: Pressure Pain Threshold
Description: Pressure pain threshold is an electronic device used to measure the amount of force that is required to produce pain when comparing baseline, week two, four and eight.
Time Frame: Pressure Pain Threshold score at week two
Measure: Mean (Standard Error); unit: pound per centimeter square
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
pound per centimeter square
  Right Pressure Pain Threshold | 4.7 (0.3) | 4.6 (0.4)
  Left Pressure Pain Threshold | 4.5 (0.3) | 4.5 (0.4)

18. Secondary Outcome: Pressure Pain Threshold
Description: as for outcome 17
Time Frame: Pressure Pain Threshold score at week four
Measure: Mean (Standard Error); unit: pound per centimeter square
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
pound per centimeter square
  Right Pressure Pain Threshold | 5.6 (0.5) | 5.3 (0.5)
  Left Pressure Pain Threshold | 5.8 (0.6) | 5.6 (0.5)

19. Secondary Outcome: Pressure Pain Threshold
Description: as for outcome 17
Time Frame: Pressure Pain Threshold score at week eight
Measure: Mean (Standard Error); unit: pound per centimeter square
Arm/Group | Combined Intervention Group | The Standard Intervention
Number analyzed (Participants) | 18 | 20
pound per centimeter square
  Right Pressure Pain Threshold | 5.8 (0.6) | 4.9 (0.4)
  Left Pressure Pain Threshold | 5.5 (0.7) | 5.4 (0.6)

ADVERSE EVENTS:
Time Frame: In the combined intervention group, one participant was excluded from the study at week two from base line measurement (second visit). Adverse events in each subject was monitored from baseline through the study completion (e.g., 8-weeks).
Description: In the combined intervention group, one participant reported a specific neck pain at week two of the study which required the patient to be excluded from the study.
Groups:
- The Combined Intervention Group: The combined intervention group: The combined intervention group received the cervical passive mobilization, stretching, and home program (Stretching and ROM exercise).
  Stretching, cervical passive mobilization, and range of motion: The manual therapy was conducted by a physical therapist who has experience in manual therapy and is licensed from the California Board of Physical Therapy. The manual therapy intervention will consist of Passive Accessory Intervertebral Movements (PAIVMs). The nature of PAIVMs techniques were selected by the physical therapist based on the participant's condition.
  Stretching exercise will be given to the participants by the physical therapist. Stretching techniques were performed in the combined intervention group for 30 seconds and repeated 3 times twice a week in the following order on the following muscles: an
- The Standard Intervention: The standard intervention: The standard intervention group received cervical mobilization and home program (ROM exercises).
  Cervical mobilization and range of motion: The manual therapy was conducted by a physical therapist who has experience in manual therapy and is licensed from the California Board of Physical Therapy. The manual therapy intervention will consist of Passive Accessory Intervertebral Movements (PAIVMs). The nature of PAIVMs techniques was selected by the physical therapist based on the participant's condition.
  Active Cervical Range of Motion Exercises (ACROM) were performed 10 repetitions 3-4 times daily. Subjects were advised to maintain their usual activity within the limits of pain. The ACROM exercise consisted of the subject placing fingers over the manubrium bone and placing chin on the fingers. The subject was then instructed to rotate to one side as f
Arm/Group | The Combined Intervention Group | The Standard Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 1/20 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Combined Intervention Group (N=20) | The Standard Intervention (N=22)
Developed specific neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — paresthesia on pinna both side L>R

LIMITATIONS AND CAVEATS:
This study had some limitations which they are short follow up period, no control group, and small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03194490/Prot_SAP_000.pdf